CLINICAL TRIAL: NCT01479959
Title: Determination of Optimal PEEP Level Under Patient Control in Tracheostomized Ventilated Patients
Brief Title: Impact of Patient Controlled Positive End-expiratory Pressure on Speech in Tracheostomized Ventilated Patients
Acronym: OptiPEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Versailles (Other)
Collaborators: Adep Assistance (Other)
Responsible Party: Principal Investigator, PRIGENT, Dr Helene PRIGENT MD, University of Versailles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Optipep -10-007
Record Dates: First submitted 2011-11-17; First posted 2011-11-28 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Respiratory Failure
Keywords: Tracheostomy; positive end expiratory pressure; speech; respiratory failure; ventilation; neuromuscular disorders
MeSH Terms: conditions — Speech; Respiratory Insufficiency; Respiratory Aspiration; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No PEEP level (Active Comparator): protocol conducted while no PEEP is applied
  Interventions: Device: Eole 3 ventilator - Resmed
- effective PEEP level (PEEPeff) (Active Comparator): PEEP level allowing the entire expiratory volume to go through the upper airways during quiet breathing
  Interventions: Device: Eole 3 ventilator - Resmed
- intermediate PEEP level (PEEP50) (Active Comparator): 50% of PEEPeff
  Interventions: Device: Eole 3 ventilator - Resmed

INTERVENTIONS:
Device: Eole 3 ventilator - Resmed — positive end expiratory pressure is added to the ventilation mode and it is activated by a switch under patient's control
  Other Names: Goodnight 420E, Tyco Healthcare, Puritan Bennett

SUMMARY:
Adequate communication is a major part of the quality of life of tracheostomized ventilator dependent patients. Maintaining speech is therefore major goal in the management of these patients.

The use of a positive end-expiratory pressure (PEEP) during ventilation has allowed the improvement of speech. The best level for speech may vary from one patient to the other The purpose of this study is to determine individually the most efficient PEEP level in terms of speech while obtaining the most secure condition and the best possible respiratory tolerance. In order to improve the latter, the investigators will use a device which allows the patients to control the activation of PEEP so that they can use it only when needed (i.e. when they wish to speak). The investigators will compare the effect of different PEEP level to try to determine the best compromise to improve speech in tracheostomized ventilator-dependent patients.

DETAILED DESCRIPTION:
Context :

Allowing a functional communication is a major issue in order to preserve quality of life in tracheostomized ventilator-dependent patients.

We showed in a previous study that the use of a positive end-expiratory pressure (PEEP) in neuromuscular tracheostomized ventilator-dependent patients improved speech as it allows the patient to expire (at least partly) through the upper airways therefore to speak during expiration. The use of PEEP has been compared to the use of a phonation valve placed on the ventilator circuit which allows a complete expiration through the upper airways and therefore speech. Both techniques seem similar in terms of efficiency on speech; PEEP, however, is better tolerated and seems to be more secure (the system remains open during expiration decreasing the risk of high pressure, it does not require any handling of the ventilator circuit).

Optimal PEEP level allowing the patient to expire the total expiratory volume through the upper airways PEEPeff may vary from one patient to the other. We seek to determine individual PEEPeff and to compare it to 50% of its value (PEEPef50). Indeed, while PEEPeff may constitute the best level for expiratory speech as it mimics the mechanisms of a phonation valve without some of its fallbacks, by preventing expiration through the expiratory circuit of the ventilator, it also may lengthen expiration, delaying inspiration which allows speech, and facilitate hyperinflation leading to respiratory discomfort as we have previously observed with some patients using a phonation valve. Optimal PEEP level would be the best compromise between best possible phonation and best possible respiratory comfort and therefore could be lower than PEEPeff.

In order to improve respiratory comfort with higher PEEP level, we developed a prototype ventilator in which PEEP is activated by a switch under the control of patients who may activate it only when needed (during speech period).

Objective :

The main objective of the study is to optimize PEEP use both by determining individually its most appropriate level and by evaluation its use overtime to allow the best possible speech with the best respiratory comfort and the most secure condition for tracheostomized ventilated patients. Different PEEP levels will be evaluated and PEEP activation will be controlled by the patients.

Methods:

Open randomized monocentric cross-over study (the patients are their own control).

Optimal PEEP level (PEEPeff), defined as PEEP-level allowing complete expiration through the upper airways, will be determined for each patient. Speech and respiratory parameters were studied without PEEP, with PEEPeff and an intermediate PEEP-level(PEEP50). Flow and airway pressure will be measure and upper airways resistance will be calculated. Microphone speech recordings were subjected to both quantitative measurements and qualitative assessments of speech.

For each PEEP level the following protocol will be conducted: 5 minutes of quiet breathing with PEEP, 10 minutes spontaneous conversation, then speech trial(maximal sustained sound, glissando, text reading).

Subjective evaluation of speech and respiratory comfort(by the patient) and objective evaluation of speech improvement according to PEEP level (reading duration, phonation duration, voice quality, assessments of speech including an intelligibility score, a perceptual score and an evaluation of prosody analyzed by two experimented speech therapists blinded to PEEP level). Evaluation of the PEEP control button use by the patient.

Inclusion criteria:

Neuromuscular adult patients, tracheotomized and on long-term ventilation with a cuffless tube, on assist-control volumetric ventilation, in stable state at the time of the study.

Number of patients, center:

Considering it is a pilot study, 14 subjects will be included for the study. The subjects will be recruited in the home ventilation unit of the intensive care department of the R. Poincare teaching hospital (Garches, France) during their usual follow-up for their chronic respiratory failure.

Duration of study: 12 months. Duration of participation for each patient will be 1h30.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Stable state upon inclusion
* Neuromuscular patients, tracheostomized and on long term ventilation with a cuffless tube
* Assist control volumetric ventilation mode
* Signed consent form

Exclusion Criteria:

* Pregnancy
* Patients unable to read
* Acute respiratory failure
* Contra-indication of PEEP use
* Lack of social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Efficiency of PEEP level on speech | 20 minutes
  Measurement of the duration of a text passage reading, the maximal phonation time throughout the repsiratory cycle.

SECONDARY OUTCOMES:
Effect of PEEP level on voice quality | 20 minutes
  Subjective evaluation by the patients with a visual analogic scale. Objective evaluation by two speech therapists (blinded to speech condition)assessing intelligibility, perceptual quality and prosody
Respiratory Comfort evaluated with a visual analogic scale by patients | 20 minutes
Respiratory tolerance | 20 minute
  Evaluation of respiratory tolerance through measurements of oxygen saturation , heart rate and respiratory rate
Use of PEEP control switch | 20 minutes
  number of use of the PEEP control switch during the text passage reading

CONTACTS AND LOCATIONS:
Overall Officials: Helene PRIGENT, MD, Principal Investigator — Hôpital Raymond Poincaré - APHP; Frederic LOFASO, MD-PhD, Study Director — University of Versailles
Locations (1):
- Hopital Raymond Poincare, Garches, France

REFERENCES:
- [Background] Prigent H, Samuel C, Louis B, Abinun MF, Zerah-Lancner F, Lejaille M, Raphael JC, Lofaso F. Comparative effects of two ventilatory modes on speech in tracheostomized patients with neuromuscular disease. Am J Respir Crit Care Med. 2003 Jan 15;167(2):114-9. doi: 10.1164/rccm.200201-026OC. Epub 2002 Oct 4. PMID 12406841
- [Background] Prigent H, Garguilo M, Pascal S, Pouplin S, Bouteille J, Lejaille M, Orlikowski D, Lofaso F. Speech effects of a speaking valve versus external PEEP in tracheostomized ventilator-dependent neuromuscular patients. Intensive Care Med. 2010 Oct;36(10):1681-1687. doi: 10.1007/s00134-010-1935-0. Epub 2010 Jun 10. PMID 20535605
- [Background] Pellegrini N, Pelletier A, Orlikowski D, Lolierou C, Ruquet M, Raphael JC, Lofaso F. Hand versus mouth for call-bell activation by DMD and Becker patients. Neuromuscul Disord. 2007 Jul;17(7):532-6. doi: 10.1016/j.nmd.2007.03.016. Epub 2007 May 29. PMID 17533130
- [Background] Bach JR, Alba AS. Tracheostomy ventilation. A study of efficacy with deflated cuffs and cuffless tubes. Chest. 1990 Mar;97(3):679-83. doi: 10.1378/chest.97.3.679. PMID 2407453
- [Background] Hoit JD, Banzett RB, Lohmeier HL, Hixon TJ, Brown R. Clinical ventilator adjustments that improve speech. Chest. 2003 Oct;124(4):1512-21. doi: 10.1378/chest.124.4.1512. PMID 14555587
- [Background] Hoit JD, Shea SA, Banzett RB. Speech production during mechanical ventilation in tracheostomized individuals. J Speech Hear Res. 1994 Feb;37(1):53-63. doi: 10.1044/jshr.3701.53. PMID 8170131
- [Derived] Garguilo M, Leroux K, Lejaille M, Pascal S, Orlikowski D, Lofaso F, Prigent H. Patient-controlled positive end-expiratory pressure with neuromuscular disease: effect on speech in patients with tracheostomy and mechanical ventilation support. Chest. 2013 May;143(5):1243-1251. doi: 10.1378/chest.12-0574. PMID 23715608